CLINICAL TRIAL: NCT05419115
Title: Use of a Novel SUBCUTaneous Preparation of Furosemide to Facilitate Early Supported Discharge of Patients With Heart Failure: a Multicentre, Phase II, Randomised, Parallel Group, Active Comparator Controlled Trial
Brief Title: Use of a Novel SUBCUTaneous Preparation of Furosemide to Facilitate Early Supported Discharge of Patients With Heart Failure
Acronym: SUBCUT-HF II
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004833-19
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: randomised, parallel-group, active comparator controlled trial
Masking Description: Not possible
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Open label, 1:1 randomisation to usual care in hospital vs early supported discharge with SQIN-Furosemide administered via SQIN-Infusor.
  Usual care: Usual care as per institutional practice (including IV diuretics)
- Early supported discharge (Experimental): Open label, 1:1 randomisation to usual care in hospital vs early supported discharge with SQIN-Furosemide administered via SQIN-Infusor.
  Early supported discharge: with SQIN-Furosemide and SQIN-Infusor. SQIN-Furosemide: 80mg of SQIN-Furosemide in each cartridge; 5 hours running time; up to 2 applications in 24h (maximum dose of 160mg of SQIN-Furosemide in 24h). SQIN-Infusor: patient/carer administered.
  Interventions: Drug: SQIN-Furosemide; Device: SQIN-Infusor

INTERVENTIONS:
Drug: SQIN-Furosemide — The investigational furosemide formulation (SQIN-Furosemide) is a Captisol®buffered solution of 80mg furosemide in 2.7 mL (30 mg/mL) at pH 7.4 (range: 7.0 to 7.8). SC infusion will be performed using the SQIN-Infusor which will deliver 2.7 mL of the SQIN-Furosemide formulation (80mg) over approximately 5 hours, using a biphasic delivery profile.
  Arms: Early supported discharge
Device: SQIN-Infusor — The investigational device (SQIN-Infusor) is an on-body delivery system that consists of a RU, DU, plus a charger (Figure 2). For the purpose of SUBCUT-HF II trial, the RU will be used for multiple infusions for a single participant. The DU will be used only once per infusion and disposed of. The RU must be charged after each use and will not restart for the next infusion without charging. Charging takes up to 15 minutes. SQIN-Infusor is a bespoke system, adapted from the design of a SC insulin pump. The RU consists of the drive-unit, the controllers, the rechargeable battery, and the user interface.
  Arms: Early supported discharge

SUMMARY:
To investigate whether an early supported discharge strategy for patients admitted to hospital because of HF, using a pH neutral subcutaneous (SC) furosemide formulation (SQINFurosemide) at home (delivered by non-CE marked SQINInfusor), compared to a usual care strategy with intravenous (IV) furosemide in hospital, results in an increased number of days spent alive and out of hospital (DAOH) at 30 days.

DETAILED DESCRIPTION:
HF is associated with frequent and lengthy hospitalisations. These hospitalisations are usually as a result of congestion, and the standard treatment of this is decongestion with intravenous (IV) diuretic (usually furosemide). This is usually delivered in a hospital setting. A new formulation of a pHneutral furosemide (SQIN-Furosemide) that can be delivered subcutaneously (SC) by a small patch pump (SQIN-Infusor) has been developed. Bioavailability of SQIN-Furosemide is similar to IV furosemide. This trial will test the efficacy and safety of novel SC furosemide 30mg/ml (SQIN-Furosemide), delivered in a home environment (compared to usual care strategy with IV furosemide delivered in secondary care) as part of a novel early supported discharge strategy in patients admitted to hospital with HF.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female ≥18 years of age
* Meet European Society of Cardiology (ESC) criteria for diagnosis of HF1

  * Elevated natriuretic peptide (BNP> 100 pg/mL or NTproBNP >300 pg/mL)
  * Signs and symptoms of HF
  * Echocardiographic structural or functional abnormality according to ESC guidelines
* Have received IV diuretic for treatment of HF within preceding 24 hours
* Be less than 96 hours after admission to hospital
* Requiring IV diuretics for a minimum of 24 hours after screening
* Have an echocardiogram or other assessment of cardiac structure and function within preceding 12 months or at screening
* Have a home environment that allows the patient to be able to mobilise within their residence and be able to pass urine into their toilet (unless catheterised)
* Able to operate (or has a caregiver who can operate) SQIN-Infusor (as assessed by training on a dummy device at screening)

Exclusion Criteria:

* Unable to consent due to significant cognitive impairment or lack of capacity
* Unable to operate SQIN-Infusor (or no caregiver who is able to operate the device)
* Geographical reasons preventing follow-up visits
* Pregnancy or breast-feeding
* Requiring treatment with IV furosemide >250 mg furosemide per day in the opinion of the treating physician
* Left sided valve disease with planned surgery or percutaneous intervention
* Type 1 myocardial infarction during index hospitalisation (participants with type 2 myocardial infarction can be included)2
* Renal impairment, defined as estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73 m 2 at screening
* Reasons (other than HF) which may prevent discharge from hospital, such as social circumstances or other significant medical condition (at investigator discretion)
* Women of childbearing potential
* Patient on active cardiac transplant waiting list
* Patient requiring on-going inotropic, vasopressor or intraaortic balloon pump support
* Potassium <3.0 mmol/L
* Potassium >6.0 mmol/L
* Sodium <125 mmol/L
* Any surgical or medical condition which, in the opinion of the investigator, may pose an undue risk to the subject, interfere with participation in the study or which may affect the integrity of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Days Alive Out of Hospital | 30 days
  Days spent alive and out of hospital (DAOH), from randomisation to 30 days.

SECONDARY OUTCOMES:
Length of index hospitalisation | 30 days
  Length of index hospitalisation
Change in quality of life | 60 days
  Change in quality of life at 60 days (assessed by Kansas City Cardiomyopathy Questionnaire [KCCQ-12]) [0-100]
Days Alive Out of Hospital | 60 days
  Days spent alive and out of hospital (DAOH), from randomisation to 60 days.
Total number of HF hospitalisations at 60 days | 60 days
  Total number of HF hospitalisations at 60 days
CV death or first HF hospitalisation at 60 days | 60 days
  CV death or first HF hospitalisation at 60 days
CV mortality at 60 days | 60 days
  CV mortality at 60 days
Safety as determined by treatment emergent adverse events (TEAEs) (including serious adverse events [SAEs]) and adverse drug events (ADEs) (including serious adverse drug events [SADEs]) | 60 days
  Safety as determined by treatment emergent adverse events (TEAEs) (including serious adverse events [SAEs]) and adverse drug events (ADEs) (including serious adverse drug events [SADEs])
Any device failures (e.g., adhesive failure and drug delivery failure) | 60 days
  Any device failures (e.g., adhesive failure and drug delivery failure)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Petrie, MBChB, Principal Investigator — University of Glasgow; Ross Campbell, MBChB, Principal Investigator — University of Glasgow
Locations (22):
- United Kingdom (22):
  - Stoke Mandeville Hospital, Aylesbury, England
  - Basildon University Hospital, Basildon, England
  - Blackpool Victoria Hospital, Blackpool, England
  - University Hospitals Dorset, Bournemouth, England
  - Southmead Hospital, Bristol, England
  - University Hospital of North Tees, Hardwick, England
  - Wycombe General Hospital, High Wycombe, England
  - Leeds General Infirmary, Leeds, England
  - Glenfield Hospital, Leicester, England
  - St Thomas' Hospital, London, England
  - St. George's University of London, London, England
  - Manchester Heart Centre, Manchester, England
  - Queen Alexandra Hospital, Portsmouth, England
  - Sunderland Royal Hospital, Sunderland, England
  - University Hospital Ayr, Ayr, Scotland
  - Ninewells Hospital, Dundee, Scotland
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Forth Valley Hospital, Larbert, Scotland
  - Queen Elizabeth University Hospital, Glasgow, Strathclyde
  - University Hospital Monklands, Airdrie
  - University Hospital Southampton, Southampton
  - The Great Western Hospital, Swindon

IPD SHARING:
Plan to Share IPD: Undecided